CLINICAL TRIAL: NCT02237872
Title: Assessment of MRI Accuracy for the Detection of Brown Adipose Tissue Using [18F]-2-fluoro-2-deoxy-D-glucose (Fluorodeoxyglucose) -PET as a Gold Standard
Brief Title: Detection of Brown Adipose Tissue by Magnetic Resonance Imaging
Acronym: BAT_PET/MRI
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 14-1980
Record Dates: First submitted 2014-09-09; First posted 2014-09-11 (Estimated); Last update posted 2025-10-01 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Brown Adipose Tissue
Keywords: Brown Adipose Tissue; MRI and PET detection of brown adipose tissue
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy volunteers exposed to cold to activate brown fat

SUMMARY:
The primary goal of this study is to assess the accuracy of conventional fat fraction proton MRI for the detection of Brown Adipose Tissue (BAT) in healthy subjects using [18F]-2-fluoro-2-deoxy-D-glucose (fluorodeoxyglucose) -PET as gold standard.

In this pilot study, MRI and PET imaging of BAT of healthy adult volunteers will be performed on a combined PET/MRI scanner under mild cold condition.

DETAILED DESCRIPTION:
In the fight against obesity, brown adipose tissue (BAT) is considered to be the newest target. The hypothesis is that this tissue is partially responsible for the imbalance between energy intake and energy expenditure that keeps lean people lean and obese people obese.

The detection of this tissue in adult humans represents an unmet need. BAT is difficult to detect and measurements of tissue fat fraction performed by magnetic resonance imaging have been proposed as a mean to differentiate the highly hydrated brown fat from the less hydrated white adipose tissue and from muscle.

To this end, the objective of this study is to assess the accuracy of magnetic resonance fat fraction measurements for the detection of BAT volume in adult humans, while using PET with fluorodeoxyglucose as gold standard.

For this study subjects will undergo a combined MRI/PET scan. The scans will be done during stimulation of thermogenic activity by mild cold exposure.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must be fully informed and have signed consent.
* BMI < 34
* Normal neurological and psychological development / able to give consent
* Willingness to participate in this study

Exclusion Criteria:

* Subjects less than 18 years of age
* Severe claustrophobia
* Women who are pregnant, nursing an infant or planning to become pregnant in the next 30 days
* People who have a condition that makes MRI unsafe for them (for example, cardiac pacemaker, epicardial pacemaker leads, cochlear implants, metal aneurysm clip, iron filings in your eyes or metal halo devices)
* Have had radiation therapy or chemotherapy in the 2 months prior to PET scan
* Subjects are taking medications that may interfere with BAT detection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult human with a BMI <28
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2015-08-27 (Actual); Study Completion 2015-08-27 (Actual)

PRIMARY OUTCOMES:
Average dice similarity coefficient | Up to 1 year after the imaging scan
  The average dice similarity coefficient will be measured to assess the overlap between MRI and PET maps

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Tamara Branca, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Biomedical Research Imaging Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided